CLINICAL TRIAL: NCT04486638
Title: Dengvaxia US Pregnancy Registry: A Surveillance Study to Assess the Safety of Dengvaxia Among Exposed Pregnant Women and Their Offsprings (DNG00044)
Brief Title: Dengvaxia US Pregnancy Registry
Acronym: DNG00044
Status: Recruiting | Type: Observational
Sponsor: Sanofi Pasteur, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Other Study IDs: DNG00044; DNG00044 (Other: Sanofi Identifier); U1111-1243-6064 (Registry Identifier: ICTRP)
Record Dates: First submitted 2020-07-22; First posted 2020-07-24 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: Dengue Virus Infection
MeSH Terms: conditions — Dengue | interventions — Dengue Vaccines

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 22 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No

GROUPS / COHORTS (1):
- Pregnant women and their offspring(s): Women and their offspring(s) exposed to Dengvaxia during pregnancy
  Interventions: Biological: Dengue Tetravalent Vaccine, Live

INTERVENTIONS:
Biological: Dengue Tetravalent Vaccine, Live — Pharmaceutical form: Powder and solvent for suspension for injection Route of administration: Subcutaneous

SUMMARY:
The primary objective of this study is to assess maternal, obstetrical, pregnancy, and neonatal and infant outcomes among women and their offspring(s) vaccinated with Dengvaxia during their pregnancy

DETAILED DESCRIPTION:
Exposed pregnant women will be followed up to the end of their pregnancy, and the offspring(s) will be followed up to 1 year of age.

ELIGIBILITY:
The eligible population will include pregnant women of any age and their offspring(s) residing in the US and its Territories whose Dengvaxia pregnancy exposure is reported to the pregnancy registry.

Reports of Dengvaxia pregnancy exposure must contain the following information to be included in the registry:

* Sufficient evidence to confirm the case qualifies as "exposed during pregnancy";
* Vaccine name (brand or generic) is provided (i.e., including manufacturer unknown exposures).

The above information is not intended to contain all considerations relevant to a patient's potential participation in a clinical trial.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Pregnant women of any age and their offspring(s) residing in the US and its Territories whose Dengvaxia pregnancy exposure is reported to the pregnancy registry
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2029-06-30 (Estimated); Study Completion 2029-06-30 (Estimated)

PRIMARY OUTCOMES:
Percentage of pregnant women with maternal adverse events | From vaccination until end of follow-up (maximum 22 months after cohort entry)
  Maternal adverse events are reported as serious or non-serious
Pecentage of women with obstetrical adverse events | From vaccination until 1 month post-delivery
  Obstetrical adverse events are collected during pregnancy, labour, delivery and puerperium, and are reported as serious or non-serious
Percentage of participants with adverse pregnancy outcome | On day of birth
  Adverse pregnancy outcomes include ectopic pregnancy, elective/induced abortion with no fetal defect(s) or fetus status unknown, elective/induced abortion with fetal defect(s), spontaneous abortion/miscarriage (<20 weeks), stillbirth/fetal death at 20-27 weeks, fetal death at ≥28 weeks, and fetal death due to maternal death
Percentage of offsprings with neonatal adverse events | From day of birth to 28 days post-birth
  Neonatal events are reported as serious or non-serious
Percentage of offsprings with infant adverse events | From 29 days to 365 days post-birth
  Infant events are reported as serious or non-serious

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (1):
- Investigational Site, San Juan, Puerto Rico

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org